CLINICAL TRIAL: NCT03927560
Title: Robotic-Assisted Percutaneous Coronary Intervention - A Safety and Effectiveness Study Applied to the Brazilian Public Health System
Brief Title: Robotic-Assisted Percutaneous Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Robotic First
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic Assisted Percutaneous Coronary Intervention (Experimental)
  Interventions: Procedure: Robotic Assisted Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Robotic Assisted Percutaneous Coronary Intervention — Robotic Assisted Percutaneous Coronary Intervention

SUMMARY:
Percutaneous coronary intervention is a safe procedure. However, its execution is manual, fully operator-dependent. The procedure is also associated with radiation exposure to patients and physicians. This study will evaluate the robotic assisted percutaneous coronary intervention as an alternative to manual operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age> = 18 years;
2. Symptomatic ischemic heart disease and / or objective evidence of myocardial ischemia with one or more target lesions;
3. Elective for percutaneous procedure (i.e. performed in a non-urgent context)
4. The target lesion (s) must be obstructive, with stenosis diameter > 50% (visual analysis);
5. The interventional planning of all target lesions should include robotic manipulation in at least one treatment, as judged by the operator;
6. Acceptable candidate for myocardial revascularization surgery.

Exclusion Criteria:

1. ST-segment elevation myocardial infarction in the last 48 hours before the index procedure;
2. Ejection fraction <30%;
3. Impaired renal function (creatinine> 2.0 mg / dL) or calculated creatinine clearance <30 ml / min;
4. Platelet count <100,000 cells / mm 3 or> 700,000 cells / mm 3;
5. Total Leucocytes count <3,000 cells / mm 3;
6. Suspected or documented active liver disease (including laboratory evidence of hepatitis);
7. Heart transplant recipient;
8. Allergies known to aspirin, clopidogrel, ticlopidine, ticagrelor, prasugrel, heparin, antiproliferative agents of the limus family, or stainless steel;
9. Patient with a life expectancy of less than 1 month;
10. Any significant medical condition that in the opinion of the investigator may interfere with the patient's ideal participation in this study;
11. Participation in other research in the last 12 months, unless there may be direct benefit to the research subject;
12. Any invasive cardiac or non-cardiac treatment scheduled within the first month after the index procedure.

Angiographic exclusion criteria

1. Need for non-robotic (i.e. manual) treatment of another injury in the index procedure or in the first month;
2. Target lesion not accessible by robotic treatment, according to the judgment of the operator;
3. Unprotected coronary artery trunk lesion (stenosis> 50%);
4. Angiographic thrombus;
5. Target lesion in surgical graft;
6. Total occlusion (TIMI 0 or 1 anterograde flow)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-06-10 (Estimated); Primary Completion 2020-02-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Procedure Complications | 1 day
  Death or non-fatal major acute complications on the target vessel (thrombosis, myocardial infarction, perforation or non-planned invasive treatment).
Procedure Success | 1 day
  Robotic Assisted Procedure Success

SECONDARY OUTCOMES:
Occurence of Major Events | 1 month
  Death, stent thrombosis, Myocardial Infarction, Stroke

IPD SHARING:
Plan to Share IPD: No